CLINICAL TRIAL: NCT06125613
Title: Influence de la kinésiophobie Sur l'excitabilité Des Connexions pariéto- Frontales au Cours d'un Mouvement de Pointage Chez l'Homme
Brief Title: Influence of Kinesiophobia on the Excitability of Connections Parieto-frontal During a Pointing Movement in Humans
Acronym: pIPS/M1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universite du Littoral Cote d'Opale (Other)
Responsible Party: Principal Investigator, Herve DEVANNE, PhD, Principal Investigator, Universite du Littoral Cote d'Opale
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2021-A02457-34
Record Dates: First submitted 2023-11-04; First posted 2023-11-09 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Kinesiophobia; Motor Coordination or Function; Developmental Disorder; Transcranial Magnetic Stimulation; Pain, Acute
Keywords: Kinesiophobia; Parietal posterior cortex; Motor Coordination or Function; Developmental Disorder; Transcranial magnetic stimulation; Pain attempt
MeSH Terms: conditions — Kinesiophobia; Developmental Disabilities; Acute Pain

STUDY DESIGN:
Intervention Model Description: Pre-post
Masking Description: A randomized number is allocated for all participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): Double pulse TMS method used to investigate the influence of the pIPS on M1 excitability. We set the ST intensity to evoke a 1mV MEP in the first dorsal interosseous muscle. The SC is applied at 90% of the MT on the pIPS. Our study involves two phases: Resting Phase: 10 single ST and 10 SC+ST doublets with a 4ms interstimulus interval. ST intensity is set to evoke a 1mV MEP, and SC is at 90% of the motor threshold. Movement Phase: Subjects perform a specific hand movement in response to colored light signals (green or red) projected on a screen. A brief but non-painful stimulus may coincide with the red signal to induce a fear response. A test stimulus (ST) or SC+ST doublet is delivered with a 500ms delay after each signal, allowing us to explore corticocortical influences during motor programming. 40 stimulations in total are delivered during this phase. Note that only 40 trials will be performed, and there will be no painful stimuli.
  Interventions: Behavioral: Experimental

INTERVENTIONS:
Behavioral: Experimental — In reality, there will not be 200 trials but 40, and no painful stimulus will be delivered. The objective is only to make the subject afraid of making a movement when the red stimulus appears, and for us to compare the situation "afraid to move" to that where there is no reason to be afraid in terms of corticocortical influences. The subject will then be invited, during the second experimental series, to perform the movements previously described. Whether the preparatory signal for movement is red or green, it will be followed with a delay of 500ms by a test stimulus alone (ST) or by a doublet of SC+ST stimulation. This stimulation will therefore occur during the motor programming period during which it has been shown in the literature that the pIPS exerts a facilitatory action on the primary motor cortex at a latency of 4 ms. In total, 10 ST and 10 SC-ST doublets will be delivered during the experimental series for each of the two colors, i.e. 40 stimulations in total.

SUMMARY:
Objective(s) of the trial: Better understand the interaction between kinesiophobia and motor control. Main objective: To measure the influence of induced kinesiophobia on functional connectivity between the posterior parieto-occipital region and the primary motor cortex in healthy subjects during a pointing task.

Secondary objectives: The secondary objectives will be 1) to verify the excitatory influence of pIPS stimulation on the excitability of M1 at rest and 2) to establish whether there is a correlation between functional connectivity and the level of kinesiophobia ( as measured by the Tampa Scale)

DETAILED DESCRIPTION:
This work will focus on a population of 30 healthy volunteer subjects who will be recruited via a posting within the Faculty of Sports Sciences of Lille, the University of Littoral Côte d'Opale and Eurasport. Compensation of 50 euros per subject is provided for participation in the study.

All these criteria will be reviewed during the visit to the clinical neurophysiology department during which each subject will be seen in an interview with a neurologist (Pr. Arnaud Delval, PU-PH of the clinical neurophysiology department of Lille University Hospital) before the start of the investigations. Explorations may be stopped at any time upon simple request from the participant. Each subject may leave the study by decision of the competent administrative authority, the promoter and the coordinating investigator but also by decision of a co-investigator or by decision of the interested party himself in accordance with the regulations and as mentioned in the consent. The data recorded in subjects who decide to leave the study will be partial and not exploitable, it will therefore be destroyed.

In this study, the impact of induced kinesiophobia on the functional connectivity between the PPC (posterior parietal cortex) and M1 (primary motor cortex) in healthy subjects during the preparatory phase of a pointing task will be assessed. Participants will undergo three transcranial magnetic stimulation (TMS) sessions.

The first session will be designed to define the optimal inter-stimulus intervals (ISIs) between both paired-pulses, with the conditioned stimulus (CS) applied to the PPC and the test stimulus (TS) applied to the M1. The second session will aim to define the optimal delay between the pointing start command (indicated by light signals) and the TS pulse over M1. The last session will determine whether a pointing start command related to a threat (indicated by a red light signal) has a different impact than a neutral pointing start command (indicated by a green light signal) on the functional connectivity between the PPC and M1.

To assess the personality of participants concerning kinesiophobia and fear-avoidance, participants will respond to two online questionnaires using RedCap, the Research Electronic Data Capture system. The questionnaires include the Tampa Scale for Kinesiophobia French version (TSK-CF) and the Fear-Avoidance Components Scale French version (FACS-Fr).

Following the completion of the questionnaires, participants will be seated comfortably in a reclining chair, with their feet resting on a footrest. The right arm will rest on a height-adjustable shelf. Electrodes for collecting electromyography (EMG) activity will be placed on the skin over the first dorsal interosseous (FDI) muscles of the right hand. This specific muscle is chosen due to its involvement in pointing tasks, and the cortical area controlling it is relatively large and easy to locate. The EMG electrodes will be connected to a recording system composed of a Digitimer D360 amplifier (UK) and a 1401 Micro MKII acquisition interface (Cambridge Electronic Design, Cambridge, UK). The data will be stored on a computer for offline analysis using Signal© software (Cambridge Electronic Design, Cambridge, UK).

Two figure-of-eight coils will be employed to induce a test stimulus (TS) and conditioning stimulus (CS). The first coil, with a 50 mm monophasic pulse, utilized for the test stimulus (TS), will be held tangentially to the skull over the left hemisphere's M1, which controls the right FDI muscle. It will be oriented at a 45° angle in the medial sagittal plane to induce an electric current oriented in the posterior to anterior direction. The test stimulus will be delivered at an intensity allowing a motor evoked potential (MEP) of 1mV to be obtained in a control situation over the spot generating the greatest MEP of the FDI muscle.

The second coil, with an 80 mm monophasic pulse, used for the conditioning stimulus (CS), will be positioned over the P3 spot of the 10/20 system, corresponding to the posterior region of the intraparietal sulcus (pIPS) of the left hemisphere. It will be held tangentially to the scalp along a parasagittal axis to enable proper placement of both coils on the same hemisphere. The conditioning stimulus will be applied on the pIPS at an intensity of 90% of the motor threshold (RMT), which corresponds to the smallest stimulation intensity that evokes 5 small responses (≥50 mV peak to peak) on the FDI muscle during a series of 10 stimulations in the subject at rest.

In this double-pulse TMS method, both coils used will be connected to stimulators, with the first coil (TS) connected to a Magstim stimulator (Whitland, UK) and the second coil (CS) connected to a Mag&More stimulator (Munich, Germany).

In the forthcoming experimental setup, investigators will arrange an environment in front of participants, incorporating four tactile light sensors (as shown in Fig. 1). The first sensor, white in color, will be positioned on a horizontal plane approximately thirty centimeters from the subject's bust, serving as the starting point for pointing tasks in sessions 2 and 3. The second sensor, also white, will be situated on an inclined plane (45°) facing the subjects, serving as the arrival point for pointing tasks in sessions 2 and 3. Adjacent to this second tactile light sensor on the inclined plane, a green light sensor on the left and a red one on the right will be placed to provide indications for the pointing task in session 3.

During the first TMS session, the focus will be on determining customized inter-stimulus intervals at rest. Building on a previous TMS paired pulse study that concentrated on the interaction between the PPC and ipsilateral M1 (25), various inter-stimulus intervals (ISIs) between CS and TS will be tested at 3, 4, 5, 6, 7, and 8 ms. Seven conditions will be randomly intermingled, including TS alone (MEP) and CS+TS (conditioned MEP for each of the six different ISIs). Eight responses will be collected for the test stimulus alone and eight responses for conditioned MEPs at each ISI.

The test stimulus will be delivered at an intensity to evoke an MEP of 1mV, and the conditioning stimulus will be delivered at an intensity of 90% of the resting motor threshold (RMT). Single pulses or doublets of stimulation will be spaced at an interval varying between 8 and 12 seconds. Measurements will be taken on each individual trial, and the mean peak-to-peak amplitude of the conditioned MEP will be expressed as a percentage of the mean peak-to-peak amplitude of the unconditioned test pulse. For the subsequent sessions, the customized optimal parameters for each participant, determined in the first session, will be used to best activate PPC-M1 interplay.

In the upcoming second TMS session, the focus will be on determining a customized delay after light signals. Participants will be instructed to wait for the first white horizontal tactile light sensor to turn on, signaling them to place their right index finger on it. After a few seconds, the green light will turn on, indicating that participants should prepare to lift their index finger to point at the second white tactile light sensor located on an inclined plane. Once the latter lights up white, participants are instructed to start the pointing task to touch it, turn it off, and then rest their right arm on the height-adjustable shelf, waiting for the first white horizontal tactile light sensor to turn on again for the next trial.

Building on a previous study focused on PPC-M1 functional connectivity during the early phase of movement planning, transcranial magnetic stimulation (TMS) will be delivered over M1 of the left hemisphere at different delays (50, 75, 100, and 125 ms) after the second white tactile light sensor located on an inclined plane turns on. Investigators will use the following parameters to best activate PPC-M1 interplay: the test stimulus (TS) delivered at an intensity to evoke a motor evoked potential (MEP) of 1mV, and in half of the experiments, a conditioning stimulus (CS) applied to the ipsilateral PPC with an intensity set at 90% of the resting motor threshold (RMT), using the customized optimal inter-stimulus interval (ISI) for each participant. Single pulses or doublets of stimulation will be spaced at an interval varying between 8 and 12 seconds.

To investigate the influence of kinesiophobia on PPC-M1 connectivity at rest, a fake electrode will be placed at the right Erb's point near the collarbone for each participant. Participants will be informed to perform the same task as before 100 times, with the random possibility of seeing either a green or red light signal appear on each trial. When the light signal is red, participants will receive a painful electric shock via the electrode on Erb's point with a 10% probability for each trial (triggered by lifting the finger from the sensor), with at least one painful electric shock guaranteed during this session. When the light signal is green, participants are assured not to receive a painful electric shock. In this session, 30 TS and 30 doublets of SC+TS stimuli will be delivered randomly, using the customized ISI for each participant. The TS will be delivered at an intensity to evoke an MEP of 1mV, and the SC will be delivered at an intensity of 90% of the RMT, with single pulses or doublets of stimulation spaced at an interval varying between 8 and 12 seconds.

In the future, there will not be 100 trials, but 60 trials, and no painful stimulus will be delivered. The objective will be solely to induce kinesiophobia when the red light appears to assess its influence on PPC-M1 connectivity between the "afraid to move" situation and the threat-free situation. The number of trials will be deliberately inflated to keep the participants alert and prevent them from assuming that they will reach the end of the session without experiencing any painful electric shock.

Following the acquisition of TMS measurements, investigators will reveal the real objective of the study, emphasizing the need to induce a fear of movement using the red-light stratagem, which falsely indicates the probability of receiving a painful electric shock. After this revelation, the experimenter will ask each participant to rate their confidence in the diagnosis (how credible the threat of receiving a painful electric shock is) as well as the fear generated by the possibility of experiencing a painful electric shock, whether it results in injury or not.

ELIGIBILITY:
Inclusion Criteria:

* Adult men and women
* Healthy subjects (who do not have self-reported neurological disorders)
* Subjects having signed informed consent (having a good command of French)
* Subjects affiliated or beneficiaries of a social security system

Exclusion Criteria:

* Psychiatric history obtained by questioning the doctor: people with mental retardation or severe impairment of cognitive, behavioral or affective functions prevents understanding the protocol and signing the informed consent
* Neurological history (epilepsy, stroke, operations performed on the brain or spinal cord and history of neurological diseases affecting motor skills and sensitivity)
* Subjects for whom we are unable to receive informed information (dementia, hearing problems, insufficient mastery of French etc.)
* Contraindications to TMS (epilepsy, intracranial metallic foreign bodies, hearing aids or cochlear implants)
* Taking psychotropic medications
* Persons under guardianship or curatorship
* Pregnant and breastfeeding women
* Subjects with a cardiac pacemaker

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-12-10 (Actual); Primary Completion 2023-03-08 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Influence of induced kinesiophobia on the functional connectivity between the posterior parieto-occipital region and the primary motor cortex in healthy subjects during a pointing task. | During TMS experiment
  We will measure the amplitude of the motor response evoked by TMS in the first dorsal interosseous muscle during simple stimulation (test stimulus or ST) of the left primary motor cortex in the area controlling the muscles of the right hand, and when the Test stimulus is preceded by a conditioning stimulus (CS) applied to the left pIPS. We will then calculate the ratio between the response obtained in the double-shock condition (SC-ST) with an interstimulus interval of 4 ms and that obtained in response to the ST alone. This will be our main judgment criterion.

SECONDARY OUTCOMES:
Excitatory influence of pIPS stimulation on M1 excitability at rest | During TMS experiment
  The influence of pIPS on M1 at rest will be evaluated in the same way as that mentioned for the main endpoint: we will measure the amplitude of the motor response evoked by TMS in the first dorsal interosseous muscle during a simple stimulation. (test stimulus or ST) of the left primary motor cortex in the area controlling the muscles of the right hand, and when the test stimulus is preceded by a conditioning stimulus (CS) applied to the left pIPS. We will then calculate the ratio between the response obtained in the double shock condition (SC-ST) with an interstimulus interval of 4 ms and that obtained in response to the ST alone. We already have used this technique in our laboratory in a previous study
Establish whether there is a correlation between functional connectivity and the level of kinesiophobia (as measured by the EKT) | Just before TMS experiment
  Kinesiophobia will be assessed using the French-Canadian version of the Tampa Kinesiophobia Questionnaire (EKT-CF). It takes the form of a 17-item self-reported questionnaire using a Likert scale ranging from 1 (strongly disagree) to 4 (strongly agree), with an acceptable degree of internal consistency (Cronbach's alpha = 0), satisfactory construct validity, high sensitivity to changes (intra-class correlation coefficient > 0.7). The total score is obtained by adding the value of the responses and is between 17 and 68. The value of 40/68 is considered the threshold value from which kinesiophobia becomes significant.

CONTACTS AND LOCATIONS:
Locations (1):
- Neurophysiologie clinique Hôpital Roger Salengro / CHU, Lille, Nord, France

IPD SHARING:
Plan to Share IPD: No